CLINICAL TRIAL: NCT02226016
Title: Quantitative Evaluation of Levator Palpebra Muscle Strength
Brief Title: Levator Muscle Strength Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, shay ofir, Investigator, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LEVATOR01
Record Dates: First submitted 2014-08-11; First posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Ptosis
Keywords: ptosis; blepharochalasis; dermatochalasis
MeSH Terms: conditions — Blepharoptosis; Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ptosis (Experimental): Device (measurement of levator strength in patients with upper lid ptosis)
  Interventions: Device: FG-5000A

INTERVENTIONS:
Device: FG-5000A — a measuring device for the assessment of levator muscle strength
  Other Names: an experimental measurinf device for a mechanical evaluation of the levator palpebra superioris muscle strength

SUMMARY:
The purpose of this study is to assess a new technique of measurement for the levator muscle.

this measurement may be applied during a clinical evaluation of eyelid malposition.

our purpose is to quantify the levator muscle strength and to corelate it to standard levator muscle strength assessment techniques routinley used in the oculoplastic clinic.

DETAILED DESCRIPTION:
This study will include patients refered to our oculoplastic department for evaluation of eyelid disorders (ptosis or eyelid malpositions due to various mechanical, muscular, neurogenic factors).

all patients will be over 21 years old, with eligibility for signing an informed concent form.

all patients will undergo a full clinical standard evaluation of eyelid malposition made as part of the routine evaluation of eyelid malpositions. as part of this evaluation- the levator muscles strength will be measured by monitoring the amount of millimeters of difference between the uper lid closed and open position (a regular technique for levator muscles assessment).

a second levator muscle strength evaluation will include the study device. this device is used for weight evaluation of objects. an object is measured by attaching it to the device with a metal hook and a string. the device is hand held.

for measurements of the upper lid force the device will be temporarily attached to the upper eyelid using a specially designed base made in the shape of the eyelid. the attachment will be using a sterile medical tape (plaster). this sterile base is attached to the outer eyelid and does not involve in any point any harm to the continuity of the skin, injections , harm or contact to the eyeball or any other parts of the eye. this base is attached from its back to a string witch attaches to the measuring device. the investigator holds the measuring device and asks the patient to open and close his eyes. the force that is generated while opening the upper lid is measured (in grams) by the device.

this evaluation will allow a unique first proper estimation of the true levator palpebra strength. it will be compared to the levators' strength as estimated using the routine techniques for assessing their efficacy.

the assessment will be made one time for each patient. after the measurement- the sterile tape will be removed and will be disposed. no further interventions will be made for each patient.

ELIGIBILITY:
Inclusion Criteria:

eligible for signing an informed concent form refered for eyelid evaluation in the oculoplastic department, Meir Mc

Exclusion Criteria:

previous eyelid surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
levator muscle strength quantified in grams using a unique measuring device. | each patient will undergo two measurments of the levator muscle strength using the study device during a single clinical evaluation. no further evaluations will be made for the same patient throughout the study.
  we aim to accurately measure the levator muscle strength in grams. the levator muscle will be noninvasively attached to the device using a string. while changing eye position from closure to opening- the force generated by the eyelid will be reflected through the string to the measuring device and will be displayed in grams. this will reflect the levator muscles strength.

SECONDARY OUTCOMES:
repeatability of the measurements | each patient will undergo two measurments of the levator muscle strength using the study device during a single clinical evaluation. no further evaluations will be made for the same patient throughout the study.
  we wish to evaluate the validity of these muscle strength assessments. for each patient two muscle measurements will be done by a single clinician. their results will be furtherly assessed for repeatability of the measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Arik Nemet, Dr, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical center, Kfar Saba, Israel, Israel